CLINICAL TRIAL: NCT04975854
Title: Virtual Reality Exposure Therapy Versus No Treatment for Acrophobia: A Randomized Controlled Trial
Brief Title: Virtual Reality Exposure Therapy for Acrophobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Responsible Party: Principal Investigator, Iveta Fajnerová, senior researcher, National Institute of Mental Health, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TL03000223-01
Record Dates: First submitted 2021-07-12; First posted 2021-07-26 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Specific Phobia; Acrophobia; Fear of Heights; Anxiety Disorders
Keywords: virtual reality exposure therapy; specific phobia; acrophobia
MeSH Terms: conditions — Phobia, Specific; Acrophobia; Anxiety Disorders | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Exposure (Experimental): Participants complete three 30-40-minute sessions of exposure administered via a virtual reality headset. The exposure involve exposure to various heights and height cues in the virtual city environment. Experimental group also attends 20-minute online information session (prerecorded video).
  Interventions: Behavioral: Exposure Therapy (Virtual Reality); Other: Information Session
- Control (Other): Control group attends a single 20-minute information session (prerecorded video) about general principles of exposure therapy and anxiety before the start of the study, but receives no exposure-based intervention.
  Interventions: Other: Information Session

INTERVENTIONS:
Behavioral: Exposure Therapy (Virtual Reality) — Virtual reality scenarios consists of increasingly intense exposures to phobic stimuli (e.g., looking over railings from various floor levels) with the support of the therapist. The goal of VRET is sufficient reduction in anxiety to allow the patients to expose themselves to heights in everyday situations.
  Arms: Virtual Reality Exposure
Other: Information Session — This includes 20-minute information session about general principles of exposure therapy before the start of the study.

SUMMARY:
The aim of this study is to examine the efficacy of virtual reality exposure therapy (VRET) as a treatment for specific phobia (acrophobia). The study will randomly assign 42 participants with acrophobia to one of two conditions: a) the experimental condition (consisting of 3 sessions of virtual reality exposure) or b) a control condition. Both groups will receive short information session about general principles of exposure therapy before the start of the study. After the end of the study, the waitlist group will be invited to attend the short version (one or two-sessions) of the VRET. Both groups will receive a final follow-up questionnaires 2 months after the last session.

ELIGIBILITY:
Inclusion Criteria:

* individual meeting ICD-10 criteria for diagnosis of specific phobia
* fluent in Czech

Exclusion Criteria:

* currently receiving psychological treatment for acrophobia
* psychotropic medication (unless on stable dosage for the previous 1 month and stabilized for the duration of the study)
* another severe mental disorder, such as bipolar disorder or psychotic disorder
* contradictions to using a virtual reality (e.g., epilepsy, balance problems)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Visual Height Intolerance Severity Scale (vHISS) | Immediately Post-Treatment (Controlling for Baseline Score)
  The vHISS is a 8-item scale assessing the severity of visual height intolerance with additional questions for diagnosing acrophobia. Raw score range from 0 to 13, where 0 = least severely affected and 13 = most severely affected.
Visual Height Intolerance Severity Scale (vHISS) | 2-months Post-Treatment (Controlling for Immediate Post-Treatment Score)
  The vHISS is a 8-item scale assessing the severity of visual height intolerance with additional questions for acrophobia.Raw score range from 0 to 13, where 0 = least severely affected and 13 = most severely affected.
Severity Measure for Specific Phobia-Adult (SMSP-A) | Immediately Post-Treatment (Controlling for Baseline Score)
  SMSP-A is a 10-item scale that assesses the severity of specific phobias in individuals aged 18 and older over the past 7 days. Items are scored on a 5-point Likert scale with item scores of 1-4 respectively indicating mild, moderate, severe and extreme severity of specific phobia related distress.
Severity Measure for Specific Phobia-Adult (SMSP-A) | 2-months Post-Treatment (Controlling for Immediate Post-Treatment Score)
  SMSP-A is a 10-item scale that assesses the severity of specific phobias in individuals aged 18 and older over the past 7 days. Items are scored on a 5-point Likert scale with item scores of 1-4 respectively indicating mild, moderate, severe and extreme severity of specific phobia related distress.
The IAPT phobia scale-avoidance | 2-Weeks In-Treatment (Controlling for Baseline Score)
  The IAPT phobia scale-avoidance is a single item from the outcome measures administered by the UK National Health Service's IAPT programme (Improving Access to Psychological Therapies). The patient is asked to rate his/her avoidance of heights in daily situations on a scale from 0 (would not avoid it) to 8 (always avoid it).
The IAPT phobia scale-avoidance | Immediately Post-Treatment (Controlling for Baseline Score)
  The IAPT phobia scale-avoidance is a single item from the outcome measures administered by the UK National Health Service's IAPT programme (Improving Access to Psychological Therapies). The patient is asked to rate his/her avoidance of heights in daily situations on a scale from 0 (would not avoid it) to 8 (always avoid it).
The IAPT phobia scale-avoidance | 2-months Post-Treatment (Controlling for Immediate Post-Treatment Score)
  The IAPT phobia scale-avoidance is a single item from the outcome measures administered by the UK National Health Service's IAPT programme (Improving Access to Psychological Therapies). The patient is asked to rate his/her avoidance of heights in daily situations on a scale from 0 (would not avoid it) to 8 (always avoid it).

SECONDARY OUTCOMES:
Six-item State-Trait Anxiety Inventory (STAI-6) | Immediately Post-Sessions
  The 6-item short form of the Spielberger State-Trait Anxiety Inventory (STAI) is used to measure self-reported symptoms of state anxiety with higher score indicating higher anxiety levels (prorated score range 20-80).
Subjective Units of Distress Scale (SUDS) | Through study completion, an average of 1 months. During In-Sessions: week 1-3 (reported repeatedly during each session in response to presented exposure situations).
  The SUDS is a visual analog scale in which the participant rates his/her anxiety/discomfort based on a range between 0 (no anxiety/discomfort) and 10 (very severe anxiety/discomfort). A SUDS rating will be collected at the end of each segment, reflecting maximum distress experienced during the interaction.
Anxiety Hierarchy | Immediately Post-Treatment (Controlling for Baseline Score)
  The patient is asked to develope a hierarchy of feared situations ranging from most-feared at the top to least-feared at the bottom. Then, he/she rates anticipated fear, anxiety or distress for each item (score 0-100 %, with higher score indicating higher anxiety) - according to how distressing they feel it would be to encounter that situation. The hierarchy is used to guide a process of VRET sessions.

OTHER OUTCOMES:
The Igroup Presence Questionnaire (IPQ) | Immediately Post-First Session
  The scale includes 3 subscales SP (spatial presence), INV (involvement) and REAL (experienced realism) with score range 0-7. Higher scores indication higher sense of presence. This measure might be positivelly associated with positive outcome.
Simulator Sickness Questionnaire (SSQ) | Immediately Post-First Session
  The scale evaluates cybersickness symptoms in three subscales: nausea (N), oculomotor disturbance (O), disorientation (D). Total simulator sickness raw score 0-48 (adjusted total score 0-180). Higher scores on each scale indicatestronger perceptions of the underlying sickness symptoms and aretherefore undesired. This measure might be negatively associated with positive outcome and sense of presence.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health, Klecany, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD (primary outcome measures) that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: IPD will be shared starting 6 month after the publication.
Access Criteria: Data access requests will be reviewed using an online form. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Derived] Francova A, Jablonska MK, Lhotska L, Husak J, Fajnerova I. Efficacy of exposure scenario in virtual reality for the treatment of acrophobia: A randomized controlled trial. J Behav Ther Exp Psychiatry. 2025 Sep;88:102035. doi: 10.1016/j.jbtep.2025.102035. Epub 2025 Mar 30. PMID 40186999